CLINICAL TRIAL: NCT03841227
Title: Effect of Transcranial Continuous Current Neuromodulation in Intrinsic Functional Brain Connectivity Assessed by Functional Magnetic Resonance Imaging (fMRI) in Fibromyalgia: A Randomized, Double-blind Controlled Trial
Brief Title: Effect of tDCS in Intrinsic Functional Brain Connectivity Assessed by Functional Magnetic Resonance in Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Wolnei Caumo, Professor at the Post-Graduation Program in Medical Sciences, Faculty of Medicine, UFRGS, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-0353
Record Dates: First submitted 2018-08-04; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; tDCS; fMRI; rs-fMRI
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active-tDCS (Active Comparator): 10 patients will receive Active-tDCS intervention (2mA, 20 min) at home.
  Interventions: Device: Active-tDCS
- Sham-tDCS (Sham Comparator): 10 patients will receive Sham-tDCS intervention (2mA, 20 min) at home.
  Interventions: Device: Sham-tDCS

INTERVENTIONS:
Device: Active-tDCS — Active home-based tDCS applied at home. 5 days a week for 4 weeks.
  Arms: Active-tDCS
Device: Sham-tDCS — Sham home-based tDCS applied at home. 5 days a week for 4 weeks.
  Arms: Sham-tDCS

SUMMARY:
Considering the central component of fibromyalgia (FM), the focus of research on current therapeutic approaches has been techniques that may modify the dysfunctional neuroplasticity process, such as transcranial direct current (tDCS) stimulation in order to counteract the dysfunction responsible for triggering and maintain the symptoms of FM. Although this technique is gaining space in research and in the clinical scenario, many questions remain to be answered, such as time of treatment, place to be stimulated and neurophysiological clarification of the mechanisms involved.

Based on the presented scenario, the present project was organized, being a double-blinded parallel randomized controlled trial with 20 female patients with FM diagnosed according to the criteria of the American Society of Rheumatology (2010 - reviewed in 2016) between 19 and 65 years of age, randomized to receive active or simulated anodic pole over the left dorsolateral prefrontal cortex (DLPFC) (10 patients in each group). Twenty 20-minute sessions, with a current intensity of 2 milliamperes, will be performed.

In order to respond to the objectives of this study, the IFC will be evaluated before and after the intervention, through rs-fMRI using seed-based correlation analysis (SCA). The investigators have a secondary objective to correlate structural connectivity through the technique of diffusion tensors imaging (DTI) with measures of pain, functional capacity, depressive symptoms and catastrophism to pain.

The hypothesis is that in FM there is a syndrome of dysfunction in basal intrinsic functional connectivity (IFC) and that the tDCS has a neuromodulatory effect capable of reducing connectivity between brain areas related to chronic pain and other neuropsychiatric components of FM, such as the ventrolateral thalamus, cortex motor, prefrontal cortex, insular cortex, hippocampus, periaqueductal gray matter, among others. The investigators believe that a higher cortico-thalamic IFC and between regions with high density of opioid receptors have a positive predictive response in the treatment of tDCS.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a syndrome that is characterized by generalized musculoskeletal pain, fatigue, unrepairable sleep, cognitive alterations, depressive and neurovegetative symptoms, whose neurobiological process is multiple and complex. Although it is of great relevance to the individual and to society, this pathology often does not receive the necessary attention by the organs that define the priorities of health care. Population prevalence, according to the criteria of the American Society of Rheumatology, reaches 5.4%, and the costs of care, taxes and early retirement due to disability are estimated at more than the US $ 29 billion per year in the United States. It is known that conventional pharmacological therapies produce insignificant responses in more than 50% of patients. It is postulated that these high rates of failure are due in part to a lack of knowledge about pathophysiological mechanisms. What is known so far is that the peripheral mechanisms contribute to the FM picture, but dysfunction in central neurobiological pathways surely commands the process, perpetuating the dysfunctional process that includes central sensitization (CS). CS comprises the symptoms of fibromyalgia syndrome that culminates in a state of hypersensitivity that expresses the imbalance of the excitation/inhibition processes that sustain this condition of non-pathological pain. Functional alterations of the motor cortex and its connections with subcortical structures that constitute the neuromatrix of pain have now been demonstrated. Functional magnetic resonance imaging (fMRI), using the resting-state fMRI (rs-fMRI) technique, has also demonstrated that high intrinsic functional connectivity (IFC) is related to pain intensity on FM.

Considering the central component of FM, the focus of research on current therapeutic approaches has been techniques that may modify the dysfunctional neuroplasticity process, such as transcranial direct current (tDCS) stimulation in order to counteract the dysfunction responsible for triggering and maintain the symptoms of FM. Although this technique is gaining space in research and in the clinical scenario, many questions remain to be answered, such as time of treatment, place to be stimulated and neurophysiological clarification of the mechanisms involved.

Based on the presented scenario, the present project was organized, being a double-blinded parallel randomized controlled trial with 20 female patients with FM diagnosed according to the criteria of the American Society of Rheumatology (2010 - reviewed in 2016) between 19 and 65 years of age, randomized to receive active or simulated anodic pole over the left dorsolateral prefrontal cortex (DLPFC) (10 patients in each group). Twenty 20 minute sessions, with a current intensity of 2 milliampere, will be performed.

In order to respond to the objectives of this study, the IFC will be evaluated before and after the intervention, through rs-fMRI using seed-based correlation analysis (SCA). The investigators have a secondary objective to correlate structural connectivity through the technique of diffusion tensors imaging (DTI) with measures of pain, functional capacity, depressive symptoms and catastrophism to pain.

The hypothesis is that in FM there is a syndrome of dysfunction in basal IFC and that the tDCS has a neuromodulatory effect capable of reducing connectivity between brain areas related to chronic pain and other neuropsychiatric components of FM, such as the ventrolateral thalamus, cortex motor, prefrontal cortex, insular cortex, hippocampus, periaqueductal gray matter, among others. The investigators believe that a higher cortico-thalamic IFC and between regions with high density of opioid receptors have a positive predictive response in the treatment of tDCS.

If the hypothesis is proven, the IFC data may serve as a biological marker associated with the perception of pain and its clinical presentation, and consequently, open the possibility of including IFC as a diagnostic parameter and therapeutic response. In addition to the possible contribution to knowledge production, this project aims to transfer the technology acquired and developed to the community, and thus benefit millions of people suffering from chronic FM pain with limited diagnostic and therapeutic perspectives, as well as extending the knowledge acquired for other neuropsychiatric disorders, such as depression.

ELIGIBILITY:
Inclusion Criteria:

* Literate
* Female, between 18 and 65 years old
* With the diagnosis of fibromyalgia according to the criteria of the American College of Rheumatology (2010-2016)
* Pain score equal to or greater than six on the Numerical Pain Scale (NPS 0-10) on most days of the last 3 months.
* Give informed consent to participate after the initial evaluation.

Exclusion Criteria:

* Living outside the city of Porto Alegre, RS, Brazil
* Pregnancy
* Severe Mental Illness
* tDCS contraindications
* Magnetic resonance imaging (MRI) contraindications

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Functional cerebral connectivity(rs-fMRI)to post-intervention rs-fMRI | 30 minutes
  Evaluation of functional cerebral connectivity using resting-state functional magnetic resonance imaging (rs-fMRI) between the change in baseline and post-intervention assessments.

SECONDARY OUTCOMES:
Structural cerebral connectivity | 30 minutes
  Evaluation of structural cerebral connectivity using diffusion tract imaging (DTI)

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (2):
- Brazil (2):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas e Porto Alegre (HCPA), Porto Alegre, Rio Grande do Sul